CLINICAL TRIAL: NCT05730231
Title: Comparison of Calorie Restriction With Early Time-restricted Eating and Calorie Restriction With Mid-day Time-restricted Eating and Daily Calorie Restriction
Brief Title: Clinical Trials of Effects of Time Restricted Eating on Health Parameters in Adults
Acronym: TRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Primorska (Other)
Responsible Party: Principal Investigator, Zala Jenko Praznikar, Associate professor, University of Primorska
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TRE_Clinical
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2024-08

CONDITIONS: Time Restricted Feeding; Overweight and Obesity; Inflammation; Hypercholesterolemia; Hypertension; Hyperglycemia; Antioxidative Stress; Metabolic Syndrome; Microbial Colonization
Keywords: time-restricted eating; calorie restriction; metabolic syndrome; overweight and obesity; dietary strategy
MeSH Terms: conditions — Intermittent Fasting; Overweight; Obesity; Inflammation; Hypercholesterolemia; Hypertension; Hyperglycemia; Metabolic Syndrome; Communicable Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Early time-restricted eating with calorie restriction (Experimental): Participants will follow calorie restriction with early day time-restricted eating protocol with three planned meals from 8:00 AM to 4:00 PM.
  Interventions: Other: Effects of calorie restriction and time-restricted eating on human health
- Mid-day time-restricted eating with calorie restriction (Experimental): Participants will follow calorie restriction with mid-day time-restricted eating protocol with three planned meals from 1:00 PM to 9:00 PM.
  Interventions: Other: Effects of calorie restriction and time-restricted eating on human health
- Daily calorie restriction (Experimental): Participants will follow daily calorie restriction protocol with three planned meals from 8:00 AM to 9:00 PM.
  Interventions: Other: Effects of calorie restriction and time-restricted eating on human health

INTERVENTIONS:
Other: Effects of calorie restriction and time-restricted eating on human health — Calorie restriction plan will be prepared for each participant. After nutritional data collection at baseline, all participant will attend educational sessions about healthy diet and beneficial effects of time-restricted eating. To estimate total energy needs, individuals' RMR will be measured from indirect calorimeter and multiplied by the appropriate factor of physical activity (from 1.3 to 1.6), and then a reduction of 200-500 kcal will be made. Macronutrient composition of the diet will be approximately 45-55% of carbohydrate, 30-35% of fat, and 15-20% of protein. 30% of daily energy intake will be consumed by breakfast, 40% by lunch and 30% by dinner. During posting participants will be allowed to consume only water and herbal infusions without added sugars or sweeteners. Dietary intake of participants will be followed during the study using a 24-h recall. Dietary data will be analysed using the Open Platform for Clinical Nutrition accessible through the website http://opkp.si/.

SUMMARY:
In a randomized controlled trial we will research the effect of calorie restriction with early and mid-day time-restricted eating (TRE) and daily calorie restriction on weight loss and human health parameters. Participants will be divided into three groups: early time-restriction group (8:00 AM to 4:00 PM), mid-day restriction group (1:00 PM to 9:00 PM) and daily calorie restriction group (8:00 AM to 9:00 PM). Participants will follow dietary strategy with three planned meals and calorie restriction. Anthropometrical and biochemical parameters will be measured at baseline, after one month, two months and at after three months of intervention. Resting metabolic rate, ultrasound scan of abdomen and ultrasound scan of carotid arteries will be measured at baseline and after three months of intervention. In addition, stool samples will be also taken at baseline and after three months of intervention.

DETAILED DESCRIPTION:
Obesity has become one of the world's most common diseases and is a major global public health challenge. Obesity contributes to an increased risk of developing various chronic diseases, such as diabetes, metabolic syndrome, hypertension, cardiovascular and kidney diseases and many others. Reducing excess body weight and improving eating habits decreases risk of disease and mortality. A lot of dietary strategies for weight loss are known and most of them are based on daily calorie restriction. Recently, an increasingly popular dietary strategy has been "time restricted eating (TRE)". In this strategy, all calorie intake is restricted within a consistent interval of less than 12 hours (4 - 10 hours). Eating window is limited to early part of the day - early TRE or mid-day TRE. Research shows that TRE has a number of beneficial effect on individuals, including weight loss, improvement of insulin sensitivity, hypercholesterolaemia, circadian rhythm of hormone secretion and other. Which TRE (early or mid-day TRE) has better health effects is still being investigated. It is also not clear how the timing, number and composition of individual meals affect on the health indicators, mentioned previously.

Therefore, the aim of our study is to evaluate and compare the effects of calorie restriction with early and mid-day time-restricted eating (TRE) and daily calorie restriction on weight loss and human health parameters in adults with at least two components of metabolic syndrome and yet not receiving any medication. The components of metabolic syndrome (lipid profile, blood pressure, anthropometry, inflammation status, glucose levels), antioxidative status, hormones (leptin, ghrelin, cortisol, insulin, adiponectin, cholecystokinin, melatonin, BDNF, IGF-1) will be measured. In addition changes in gene expression of different proteins will be examined. Moreover, stool samples will be also taken at baseline and after three months of intervention.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25-35 kg/m2

  + one of the following criteria:
* Increased waist circumference ≥ 94 cm in men and ≥ 80 cm in women
* Fasting plasma glucose > 5,6 mmol/L
* Elevated fasting plasma triglycerides 1,7 mmol/l
* Reduced high-density lipoprotein (HDL)-cholesterol < 1,0 mmol/l for men, < 1,3 mmol/l for women
* Elevated blood pressure, systolic blood pressure > 130 mm Hg and diastolic blood pressure > 85 mm Hg
* Without medicals for hypertension and hypercholesterolemia
* Morning or afternoon working time

Exclusion Criteria:

* Pregnant or plan to be become pregnant
* Lactating women
* Active smoking
* Diagnosis of diabetes
* Eating disorders
* Currently enrolled in a weight-management program
* Uncontrolled medical condition due to gastrointestinal, psychiatric, rheumatologic, oncologic, hematologic or endocrine diseases
* History of tumor
* History of serious cardiovascular or cerebrovascular diseases
* Taking medicines that may affect weight and appetite

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2023-03-03 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Body Weight | three months
  Changes in body weight (in kilograms) from baseline to week twelve measured with bioelectrical impedance analysis (BIA) Tanita MC-980MA

SECONDARY OUTCOMES:
Change in Body Fat | three months
  Changes in percentage of body fat from baseline to week twelve measured with bioelectrical impedance analysis (BIA) Tanita MC-980MA
Changes in Visceral Fat Rating | three months
  Changes in visceral fat rating (index) from baseline to week twelve measured with bioelectrical impedance analysis (BIA) Tanita MC-980MA. The range of the visceral fat rating (scale) is from 0 to 30. Higher scores indicate excess visceral fat (a worse outcome).
Changes in Muscle mass | three months
  Changes in muscle mass (in kilograms) from baseline to week twelve measured with bioelectrical impedance analysis (BIA) Tanita MC-980MA
LDL Cholesterol | three months
  Changes in LDL cholesterol measured by biochemical analyzer Cobass
Inflammation | three months
  Changes in C-reactive protein levels measured by biochemical analyzer Cobass
Glucose levels | three months
  Changes in glucose levels measured by biochemical analyzer Cobass
Resting metabolic rate | three months
  Changes in resting metabolic rate measured by (MedGem® Microlife, Medical Home Solutions, Inc., Golden, CO)
ultrasound scan of abdomen | three months
  ultrasound scan of abdomen measured by Resona 7 Mindray
ultrasound scan of carotid arteries | three months
  ultrasound scan of carotid arteries measured by Resona 7 Mindray
Antioxidative potential | three months
  Antioxidative potential will be determined with DPPH radical measurement.
Blood Pressure | three months
  Changes in systolic blood pressure measured by blood pressure device (Omron M3)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Primorska, Faculty of Health Sciences, Izola, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Manoogian ENC, Chow LS, Taub PR, Laferrere B, Panda S. Time-restricted Eating for the Prevention and Management of Metabolic Diseases. Endocr Rev. 2022 Mar 9;43(2):405-436. doi: 10.1210/endrev/bnab027. PMID 34550357
- [Background] Liu D, Huang Y, Huang C, Yang S, Wei X, Zhang P, Guo D, Lin J, Xu B, Li C, He H, He J, Liu S, Shi L, Xue Y, Zhang H. Calorie Restriction with or without Time-Restricted Eating in Weight Loss. N Engl J Med. 2022 Apr 21;386(16):1495-1504. doi: 10.1056/NEJMoa2114833. PMID 35443107
- [Background] Swiatkiewicz I, Mila-Kierzenkowska C, Wozniak A, Szewczyk-Golec K, Nuszkiewicz J, Wroblewska J, Rajewski P, Eussen SJPM, Faerch K, Manoogian ENC, Panda S, Taub PR. Pilot Clinical Trial of Time-Restricted Eating in Patients with Metabolic Syndrome. Nutrients. 2021 Jan 24;13(2):346. doi: 10.3390/nu13020346. PMID 33498955
- [Background] Zhang LM, Liu Z, Wang JQ, Li RQ, Ren JY, Gao X, Lv SS, Liang LY, Zhang F, Yin BW, Sun Y, Tian H, Zhu HC, Zhou YT, Ma YX. Randomized controlled trial for time-restricted eating in overweight and obese young adults. iScience. 2022 Aug 5;25(9):104870. doi: 10.1016/j.isci.2022.104870. eCollection 2022 Sep 16. PMID 36034217
- [Derived] Cresnovar T, Habe B, Mohorko N, Kenig S, Jenko Praznikar Z, Petelin A. Early time-restricted eating with energy restriction has a better effect on body fat mass, diastolic blood pressure, metabolic age and fasting glucose compared to late time-restricted eating with energy restriction and/or energy restriction alone: A 3-month randomized clinical trial. Clin Nutr. 2025 Jun;49:57-68. doi: 10.1016/j.clnu.2025.04.001. Epub 2025 Apr 8. PMID 40250088